CLINICAL TRIAL: NCT01944618
Title: forREAL: FORXIGA (DAPAGLIFLOZIN PROPANEDIOL MONOHYDRATE) PRESCRIPTION EVENT MONITORING PROGRAM
Brief Title: forREAL: FORXIGA PRESCRIPTION EVENT MONITORING PROGRAM (PEMP)
Acronym: forREAL
Status: Terminated | Type: Observational
Why Stopped: Participant Data obtained to 30Sep2015:
  Baseline data: 447 6 month data: 253 Program terminated: recruitment target not met. No analysis will be provided.
Sponsor: AstraZeneca (Industry)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: MB102-209
Record Dates: First submitted 2013-09-13; First posted 2013-09-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- T2DM patients newly prescribed Forxiga: A post-marketing evaluation of the safety of Forxiga (10 mg tablets, orally once daily for 6 months) through an observational prescription adverse event monitoring program (registry-based monitoring program) is warranted to assess real-world incidence of adverse events in routine clinical practice.
  Interventions: Drug: Forxiga

INTERVENTIONS:
Drug: Forxiga — FORXIGA is a prescription medicine used with diet, exercise and sometimes other medicines (which may include metformin; insulin; a sulfonylurea medicine such as gliclazide, glimepiride and glibenclamide; or a dipeptidyl peptidase-4 inhibitor [DPP 4 inhibitor] such as sitagliptin or saxagliptin) to control the levels of blood sugar (glucose) in patients with type 2 diabetes mellitus.
  Other Names: Dapagliflozin

SUMMARY:
The study purpose is to assess adverse events in patients with Type 2 diabetes who have newly been prescribed Forxiga for the management of glycemic control

DETAILED DESCRIPTION:
Observational Model: Other: A post-marketing evaluation of the safety of Forxiga through an observational prescription adverse event monitoring program (registry-based monitoring program) is warranted to assess real-world incidence of adverse events in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

Patients with Type 2 Diabetes who are:

* Prescribed Forxiga for glycaemic management AND
* Who have the ability to provide informed consent

Exclusion Criteria:

Patients with whom use of Forxiga is contraindicated:

* Patients with Type 1 Diabetes
* Patients with moderate to severe renal impairment [Creatinine clearance (CrCl) <60 mL/min or estimated glomerular filtration rate (eGFR) <60mL/min/1.73m²]

Additional exclusion criteria:

* Age >75 years
* Concomitant use of loop diuretics or pioglitazone
* Patients who are currently on another SGLT2 inhibitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes whom the Healthcare professional (HCP) would consider as suitable candidates for Forxiga treatment will be invited to participate in the program during routine clinical assessment
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence rates of adverse events, specifically genital infections, urinary tract infections, increased haematocrit, renal impairment, hepatic impairment, bone fractures and cancers, in particular breast, bladder, and prostate cancers | Up to 6 months
  Assessed in patients with Type 2 diabetes who are treated with Forxiga in routine Australian clinical practice
Any early adverse effects as a result of drug interactions in patients with Type 2 diabetes who are treated with Forxiga in routine Australian clinical practice | Up to 6 months
Incidence rates of spontaneously reported hypoglycaemia in patients with Type 2 diabetes who are treated with Forxiga in routine Australian clinical practice | Up to 6 months

SECONDARY OUTCOMES:
Rate of prescribing of Forxiga after its introduction to routine Australian clinical practice | Upto 6 months
Indication for prescription of Forxiga in routine Australian clinical practice | Upto 6 months
Change in efficacy and safety variables after treatment with Forxiga for at least 3 months | Baseline and 3 months
  Including:
  * HbA1c
  * Weight
  * Systolic blood pressure
  * Diastolic blood pressure
  * Heart rate
  * Serum creatinine
  * Estimated glomerular filtration rate
  * Liver function tests [Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), or bilirubin]
Subgroup analyses may be conducted for selected safety parameters | Upto 6 months
  Subgroups to be evaluated will include gender, age, diabetes duration, concomitant medication, past medical history, and measured laboratory variables (if available)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Zoungas, Professor, Study Director — Monash University; Christopher Reid, Professor, Study Director — Monash University
Locations (1):
- Local Institution, Clayton, Victoria, Australia